CLINICAL TRIAL: NCT01192295
Title: An Open-label, Multicenter Study of the Safety of Twice Daily Oxycodone Hydrochloride Controlled-release Tablets in Opioid Experienced Children From Ages 6 to 16 Years Old, Inclusive, With Moderate to Severe Malignant and/or Nonmalignant Pain Requiring Opioid Analgesics
Brief Title: Safety of Twice Daily Oxycodone Hydrochloride Controlled-release Tablets in Children With Moderate to Severe Malignant and/ or Nonmalignant Pain Requiring Opioids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTR3001; 2010-020471-23 (EudraCT Number)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2015-02-06 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pain
Keywords: Malignant pain; Nonmalignant pain; Pediatric; Opioid; Moderate to severe malignant or nonmalignant pain
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxycodone HCl controlled-release (Experimental): Oxycodone hydrochloride (HCl) controlled-release (CR)
  Interventions: Drug: Oxycodone HCl controlled-release tablets

INTERVENTIONS:
Drug: Oxycodone HCl controlled-release tablets — Oxycodone HCl controlled-release tablets at strengths of 10, 15, 20, 30, or 40 mg (20 mg - 240 mg daily) every 12 hours.
  Other Names: OxyContin

SUMMARY:
The purpose of this study is to characterize the safety of oxycodone hydrochloride (HCl) controlled-release (CR) tablets in opioid tolerant pediatric patients aged 6 to 16 years, inclusive, with moderate to severe malignant and/or nonmalignant pain requiring opioid therapy.

ELIGIBILITY:
Inclusion Criteria include:

* Male and female patients aged 6 to 16 years, inclusive, who are expected to require ongoing around-the-clock opioid treatment equivalent to at least 20-mg daily dose of oxycodone for at least 2 weeks for management of moderate to severe (based on the investigator's judgment) malignant or nonmalignant pain.
* Patients must be opioid tolerant, ie, have been treated with opioids for at least the 5 consecutive days prior to dosing and with at least 20 mg daily of oxycodone or the equivalent during at least the last 48 hours prior to the start of study drug dosing and have tolerated the therapy, as demonstrated at the start of study drug dosing.
* Patients who are currently using transdermal fentanyl should have been on the patch for at least 3 days before removing the patch and oxycodone hydrochloride (HCl) controlled-release (CR) treatment can only be initiated at least 18 hours following the removal of the transdermal fentanyl patch.
* Patients must not require more than a 240-mg total daily dose of oxycodone HCl CR tablets.
* Patients must be willing and able to swallow the oxycodone HCl CR tablets whole.
* Patients must not be currently on an investigational medication/therapy at the start of screening or during the study.

Exclusion Criteria include:

* Female patients who are pregnant or lactating.
* Patients who are allergic to oxycodone or have a history of allergies to other opioids (this criterion does not include patients who have experienced common opioid side effects [eg, nausea, constipation]).
* Patients who have received epidural opioids < 2 hours prior to the first dose of study drug or who have received epidural morphine < 12 hours prior to the first dose of study drug.
* Patients who are contraindicated for the use of opioids.
* Patients who are contraindicated for blood sampling.
* Patients who are currently being maintained on methadone for pain.
* Patients who have any planned surgery during the course of the study, with the exception of the placement of central or peripheral venous access devices.
* Patients who have had surgery within 5 days prior to Day 1 (day of first dose of study drug).
* Patients who, in the investigator's opinion, have an underlying gastrointestinal condition or other disorder that may predispose them to obstruction.

Other protocol-specific inclusion/exclusion criteria may apply.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (35):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of South Alabama, Children's and Women's Hospital, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - LS Packard Children's Hospital, Palo Alto, California
  - Bayview Research Group, LLC, Paramount, California
  - Shriners Hospitals for Children Northern California, Sacramento, California
  - The Children's Hospital, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Memorial Regional Hospital, Hollywood, Florida
  - Jackson Memorial Hospital/University of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - St. John's Mercy Medical Center, St Louis, Missouri
  - New York University Langone Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Presbyterian Blume Pediatric Hematology and Oncology Clinic, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Department of Pediatrics, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Children's Hospital at OUMC, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Ctr of Dallas, Dallas, Texas
  - Research Facility, The Woodlands, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Pediatric Hematology and Oncology, Virginia Commonwealth University Health System, Richmond, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Greece (2):
  - Agia Sophia Children's Hospital, Athens
  - Aglaia Kyriakou - Elpida Children's Oncology Unit, Athens
- Semmelweis Egyetem, II. sz. Gyermekgyogyaszati Klinika, Budapest, Hungary
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Mayer Children Hospital, Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Ein Kerem, Jerusalem
  - Schneider Children Medical Center of Israel, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Starship Children's Health, Grafton, Auckland, New Zealand
- Spitalul Clinic Judetean de Urgenta Targu Mures, Clinica pediatrie I, Târgu Mureş, Romania
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
- Sheffield Children's Hospital, Sheffield, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit: 28-Feb-2011; Last Patient Last Visit: 29-Jul-2014. The study was conducted at medical/research sites in the United States, Spain, United Kingdom, Greece, Guatemala, Hungary, Israel, and New Zealand
Groups:
- 6 to < 12 Years: Children 6 to < 12 years of age
- ≥ 12 to ≤ 16 Years: Children ≥ 12 to ≤ 16 years of age
Period: Overall Study
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Started | 27 | 128
Completed | 17 | 105
Not Completed | 10 | 23
Not completed — Adverse Event | 3 | 7
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 5
Not completed — Administrative | 4 | 6

BASELINE CHARACTERISTICS:
Population: The safety population was the group of patients who received at least 1 dose of study drug during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years | Total
Number analyzed (Participants) | 27 | 128 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.6 (1.65) | 14.5 (1.34) | 13.7 (2.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 75 | 89
  Male | 13 | 53 | 66
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 88 | 108
  Black or African American | 7 | 31 | 38
  Asian | 0 | 1 | 1
  Other | 0 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events as a Measure of Safety.
Description: Safety assessments consisted of reports of AEs, physical examinations, clinical laboratory test results, vital signs measurements, pulse oximetry (SpO2), and somnolence assessments. Safety variables were summarized descriptively within age group for the safety population.
Time Frame: Up to 4 weeks (during the study) and 7-10 days poststudy (safety follow-up assessment).
Population: The safety population was the group of patients who received at least 1 dose of study drug during the study.
Measure: Number; unit: participants
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Number analyzed (Participants) | 27 | 128
participants
  Serious adverse events | 5 | 22
  All other adverse events in ≥ 5% of patients | 13 | 60

2. Secondary Outcome: Pain Right Now Assessment by Patients Aged 6 to < 12 Years
Description: Pain right now was assessed by patients aged 6 to <12 years using the Faces of Pain Scale-Revised (FPS-R). The FPS-R is a horizontal row of 6 faces representing pain intensity, with "no hurt" at the far left and "hurts worst" at the far right; the 6 intensities are scored as 0, 2, 4, 6, 8, or 10 (the patient was not shown the numbers associated with the faces). A score of 0 means no pain, and a 10 means very much pain. Pain right now was assessed by the patient at screening; after the first dose; and, thereafter, twice daily during the AM and PM, approximately at the time of each (morning and evening) dose of oxycodone HCl CR tablets during the study treatment.
Time Frame: Baseline to week 4
Population: The safety population was the group of patients who received at least 1 dose of study drug during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 to < 12 Years
Number analyzed (Participants) | 27
units on a scale
  Baseline | 4.44 (3.250)
  Average during week 1: morning: number analyzed (Participants) | 25
  Average during week 1: morning | 4.11 (2.674)
  Average during week 1: evening: number analyzed (Participants) | 26
  Average during week 1: evening | 4.07 (2.695)
  Average during week 2: morning: number analyzed (Participants) | 23
  Average during week 2: morning | 3.66 (2.640)
  Average during week 2: evening: number analyzed (Participants) | 22
  Average during week 2: evening | 3.70 (2.686)
  Average during week 3: morning: number analyzed (Participants) | 17
  Average during week 3: morning | 3.64 (2.579)
  Average during week 3: evening: number analyzed (Participants) | 17
  Average during week 3: evening | 3.76 (2.669)
  Average during week 4: morning: number analyzed (Participants) | 14
  Average during week 4: morning | 3.13 (2.569)
  Average during week 4: evening: number analyzed (Participants) | 14
  Average during week 4: evening | 3.42 (2.974)

3. Secondary Outcome: Pain Right Now Assessment by Patients Aged ≥ 12 to ≤ 16 Years
Description: Pain right now was assessed by patients aged ≥ 12 to ≤ 16 years using the 100-mm visual analogue scale (VAS). The 100-mm VAS is a 100-mm line with 1 end marked "no pain" and the opposite end marked as "pain as bad as it could be." The patient was asked to make a mark on that line indicating his or her level of pain. The pain right now 100-mm VAS score was defined as the distance (in mm) from the "no pain" end to the patient's mark. The scale is measured on a 100 mm line: a 0 means no pain and bigger numbers indicate more pain. Pain right now was assessed by the patient at screening; after the first dose; and, thereafter, twice daily during the AM and PM, approximately at the time of each (morning and evening) dose of oxycodone HCl CR tablets during the study treatment.
Time Frame: Baseline to week 4
Population: The safety population was the group of patients who received at least 1 dose of study drug during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ≥ 12 to ≤ 16 Years
Number analyzed (Participants) | 128
units on a scale
  Baseline: number analyzed (Participants) | 126
  Baseline | 44.58 (28.291)
  Average during week 1: morning: number analyzed (Participants) | 124
  Average during week 1: morning | 40.38 (24.402)
  Average during week 1: evening: number analyzed (Participants) | 124
  Average during week 1: evening | 39.24 (23.301)
  Average during week 2: morning: number analyzed (Participants) | 122
  Average during week 2: morning | 34.49 (24.980)
  Average during week 2: evening: number analyzed (Participants) | 122
  Average during week 2: evening | 33.04 (24.778)
  Average during week 3: morning: number analyzed (Participants) | 101
  Average during week 3: morning | 32.56 (25.802)
  Average during week 3: evening: number analyzed (Participants) | 88
  Average during week 3: evening | 33.46 (24.639)
  Average during week 4: morning: number analyzed (Participants) | 53
  Average during week 4: morning | 35.58 (27.177)
  Average during week 4: evening: number analyzed (Participants) | 50
  Average during week 4: evening | 35.30 (26.711)

4. Secondary Outcome: Use of Supplemental Pain Medication
Description: Supplemental opioid and nonopioid pain medications were permitted during the study as deemed appropriate by the investigator. The dose of supplemental analgesic medication allowed was at the discretion of the investigator and within appropriate dose ranges for age and weight.
Time Frame: Baseline to week 4
Population: The safety population was the group of patients who received at least 1 dose of study drug during the study.
Measure: Number; unit: participants
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Number analyzed (Participants) | 27 | 128
participants
  Any supplemental pain medication | 24 | 112
  Any opioid supplemental pain medication | 21 | 93
  Any nonopioid supplemental pain medication | 17 | 75

5. Secondary Outcome: Parent/ Caregiver-Assessed Global Impression of Change (PGIC)
Description: The PGIC rating score variable was collected on a 7-point scale ranging from 1 to 7 (where 1 = very much improved; and 7 = very much worse). The PGIC is designed to assess overall satisfaction with the treatment. The number and percent of parent/caregivers reporting each category of PGIC response at the final visit was summarized for the safety population within age group.
Time Frame: Baseline to week 4 or early discontinuation
Population: The safety population was the group of patients who received at least 1 dose of study drug during the study.
Measure: Number; unit: participants
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Number analyzed (Participants) | 25 | 115
participants
  1 = Very much improved | 10 | 42
  2 = Much improved | 8 | 51
  3 = Minimally improved | 3 | 15
  4 = No change | 3 | 5
  5 = Minimally worse | 0 | 1
  6 = Much worse | 0 | 0
  7 = Very much worse | 1 | 1

6. Secondary Outcome: Parent/ Caregiver Assessed Functional Disability Inventory (FDI) for Patients Aged 6 to < 12 Years
Description: The FDI is a validated tool used to evaluate the degree to which children have reduced physical and psychosocial functioning because of their pain difficulties in the previous 2 weeks. The FDI comprises 15 items. Responses to each item were scored using a 5-point Likert scale. The individual scores are: (0) no trouble, (1) a little trouble, (2) some trouble, (3) a lot of trouble, and (4) impossible. A total score (ranging from 0 to 60) for the 15 items was calculated, with lower scores indicating less functional disability. The FDI was performed by the parent/ caregiver.
Time Frame: Baseline to week 4
Population: The safety population was the group of patients who received at least 1 dose of study drug during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 6 to < 12 Years
Number analyzed (Participants) | 27
units on a scale
  Baseline: number analyzed (Participants) | 26
  Baseline | 27.1 (13.06)
  Week 4: number analyzed (Participants) | 25
  Week 4 | 23.0 (13.32)

7. Secondary Outcome: Parent/ Caregiver Assessed Functional Disability Inventory (FDI) for Patients Aged ≥ 12 to ≤ 16 Years
Description: as for outcome 6
Time Frame: Baseline to week 4
Population: The safety population was the group of patients who received at least 1 dose of study drug during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ≥ 12 to ≤ 16 Years
Number analyzed (Participants) | 128
units on a scale
  Baseline: number analyzed (Participants) | 127
  Baseline | 23.2 (17.47)
  Week 4: number analyzed (Participants) | 119
  Week 4 | 20.4 (12.65)

8. Secondary Outcome: Pharmacokinetics (PK) Data of Oxycodone Hydrochloride Controlled-release Tablets
Description: A population PK analysis using sparse plasma concentration data in pediatric patients was conducted. Empirical Bayes estimates were used to calculate individual PK parameters. PK parameters were calculated and reported for each individual patient's first and last dose. Cmax was taken as the maximum simulated oxycodone concentration over the dosing interval and Cmin was the simulated oxycodone concentration when time was equal to 12 hours. Steady-state Cmin and Cmax were derived from the accumulation ratio.
  The following PK parameters are presented: Cmin / Cmax (minimum / maximum concentration); Cmin,ss / Cmax,ss (Cmin / Cmax at steady state); CAVGss (average concentration at steady state).
Time Frame: Day 1 - first dose [2-4 hrs post dose and 4-6 hrs post dose], week 4 - last dose [at pre-dose and at 2-4 hrs post dose]
Population: Full analysis population for PK consisted of patients who received at least 1 dose of study drug and had at least 1 valid PK concentration.
Measure: Median (90% Confidence Interval); unit: ng/mL
Groups:
- 6 to 16 Years: Children 6 to 16 years of age
Arm/Group | 6 to 16 Years
Number analyzed (Participants) | 105
ng/mL
  Cmin - first dose: number analyzed (Participants) | 99
  Cmin - first dose | 6.86 [2.69 to 23.1]
  Cmin - last dose: number analyzed (Participants) | 90
  Cmin - last dose | 6.35 [2.34 to 22.0]
  Cmin,ss - first dose: number analyzed (Participants) | 99
  Cmin,ss - first dose | 7.73 [2.9 to 28.8]
  Cmin,ss - last dose: number analyzed (Participants) | 90
  Cmin,ss - last dose | 7.46 [2.47 to 28.9]
  Cmax - first dose: number analyzed (Participants) | 99
  Cmax - first dose | 16.3 [7.82 to 58.2]
  Cmax - last dose: number analyzed (Participants) | 90
  Cmax - last dose | 15.8 [7.87 to 59.5]
  Cmax,ss - first dose: number analyzed (Participants) | 99
  Cmax,ss - first dose | 20.9 [9.23 to 66.1]
  Cmax,ss - last dose: number analyzed (Participants) | 90
  Cmax,ss - last dose | 17.9 [9.46 to 68.4]
  CAVGss - first dose: number analyzed (Participants) | 99
  CAVGss - first dose | 16.1 [6.84 to 53.7]
  CAVGss - last dose: number analyzed (Participants) | 90
  CAVGss - last dose | 15.7 [6.77 to 58.9]

9. Secondary Outcome: Pharmacokinetics (PK) Data of Oxycodone Hydrochloride Controlled-release Tablets - AUCtau and AUCss
Description: A population PK analysis using sparse plasma concentration data in pediatric patients was conducted. Empirical Bayes estimates were used to calculate individual PK parameters. PK parameters were calculated and reported for each individual patient's first and last dose. First-dose area under the concentration-time curve (AUC) was derived from the accumulation ratio. For all calculations, the dosing interval was assumed to be 12 hours.
  The following PK parameters are presented: AUCtau (area under the concentration-time curve from time zero to time equal to dosing interval); AUCss (AUC at steady state).
Time Frame: Day 1 - first dose [2-4 hrs post dose and 4-6 hrs post dose], week 4 - last dose [at pre-dose and at 2-4 hrs post dose]
Population: as for outcome 8
Measure: Median (90% Confidence Interval); unit: ng*hour/mL
Arm/Group | 6 to 16 Years
Number analyzed (Participants) | 105
ng*hour/mL
  AUCtau - first dose: number analyzed (Participants) | 99
  AUCtau - first dose | 181 [74.2 to 562]
  AUCtau - last dose: number analyzed (Participants) | 90
  AUCtau - last dose | 158 [77.2 to 545]
  AUCss - first dose: number analyzed (Participants) | 99
  AUCss - first dose | 194 [82.1 to 645]
  AUCss - last dose: number analyzed (Participants) | 90
  AUCss - last dose | 188 [81.3 to 707]

10. Secondary Outcome: Pharmacokinetics (PK) Data of Oxycodone Hydrochloride Controlled-release Tablets - Time to Maximum Concentration (Tmax)
Description: A population PK analysis using sparse plasma concentration data in pediatric patients was conducted. Empirical Bayes estimates were used to calculate individual PK parameters. PK parameters were calculated and reported for each individual patient's first and last dose.
Time Frame: Day 1 - first dose [2-4 hrs post dose and 4-6 hrs post dose], week 4 - last dose [at pre-dose and at 2-4 hrs post dose]
Population: as for outcome 8
Measure: Median (90% Confidence Interval); unit: Hours
Arm/Group | 6 to 16 Years
Number analyzed (Participants) | 105
Hours
  Tmax - first dose: number analyzed (Participants) | 99
  Tmax - first dose | 3.75 [2.5 to 5.75]
  Tmax - last dose: number analyzed (Participants) | 90
  Tmax - last dose | 3.75 [2.5 to 5.75]

11. Secondary Outcome: Pharmacokinetics (PK) Data of Oxycodone Hydrochloride Controlled-release Tablets - Accumulation Ratio
Description: A population PK analysis using sparse plasma concentration data in pediatric patients was conducted. Empirical Bayes estimates were used to calculate individual PK parameters. PK parameters were calculated and reported for each individual patient's first and last dose. The accumulation ratio is used to derive steady-state Cmin and Cmax and first-dose area under the concentration-time curve (AUCtau).
Time Frame: Day 1 - first dose [2-4 hrs post dose and 4-6 hrs post dose], week 4 - last dose [at pre-dose and at 2-4 hrs post dose]
Population: as for outcome 8
Measure: Median (90% Confidence Interval); unit: Ratio
Arm/Group | 6 to 16 Years
Number analyzed (Participants) | 105
Ratio
  Accumulation ratio - first dose: number analyzed (Participants) | 99
  Accumulation ratio - first dose | 1.14 [1.03 to 1.40]
  Accumulation ratio - last dose: number analyzed (Participants) | 90
  Accumulation ratio - last dose | 1.14 [1.03 to 1.42]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported from start of study participation through the period beyond study completion.
Description: AEs were learned of through spontaneous reports and/or patient interview, or were observed during physical examinations or other safety assessments. Ongoing AEs were followed until resolution or 30 days after last study drug dose. Serious AEs up to 30 days following the last study visit were followed until the AE or sequelae resolved or stabilized.
Arm/Group | 6 to < 12 Years | ≥ 12 to ≤ 16 Years
Serious Adverse Events (participants affected / at risk) | 5/27 | 22/128
Other Adverse Events (participants affected / at risk) | 13/27 | 60/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 6 to < 12 Years (N=27) | ≥ 12 to ≤ 16 Years (N=128)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 — Outcome: Death
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 2 | 5
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — Outcome: Death
Balance disorder (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 1 — Outcome: Death. 1 patient (6 to < 12 Years) experienced 3 serious AEs resulting in death: coma, convulsion, and respiratory disorder; 1 patient (≥ 12 to ≤ 16 Years) experienced 2 serious AEs resulting in death: coma and hypoxia.
Convulsion (Nervous system disorders) | 1 | 0 — Outcome: Death. 1 patient (6 to < 12 Years) experienced 3 serious AEs resulting in death: coma, convulsion, and respiratory disorder.
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 0 | 1
Status migrainosus (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Outcome: death. 1 patient (≥ 12 to ≤ 16 Years) experienced 2 serious AEs resulting in death: coma and hypoxia.
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — 1 patient (6 to < 12 Years) experienced 3 serious AEs resulting in death: coma, convulsion, and respiratory disorder.
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6 to < 12 Years (N=27) | ≥ 12 to ≤ 16 Years (N=128)
Vomiting (Gastrointestinal disorders) | 6 | 26
Nausea (Gastrointestinal disorders) | 3 | 20
Constipation (Gastrointestinal disorders) | 4 | 12
Pyrexia (General disorders) | 5 | 8
Headache (Nervous system disorders) | 3 | 17
Dizziness (Nervous system disorders) | 0 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days